CLINICAL TRIAL: NCT03537911
Title: Cognitive Support Program for Patients With Brain Metastases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 16-6056
Record Dates: First submitted 2018-04-21; First posted 2018-05-25 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Metastases, CNS
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cognitive Support Program (Experimental): Three individual sessions of supportive psychoeducation, mindfulness practice, and strategy training (e.g., strategies to improve memory or concentration), with practice applying program content between sessions.
  Interventions: Behavioral: Cognitive Support Program

INTERVENTIONS:
Behavioral: Cognitive Support Program — Three individual sessions of supportive psychoeducation, mindfulness practice, and strategy training (e.g., strategies to improve memory or concentration), with practice applying program content between sessions.

SUMMARY:
This study evaluates the feasibility and preliminary efficacy of a brief cognitive-behavioural program designed to improve cognitive functioning in people with brain metastases.

DETAILED DESCRIPTION:
Cognitive impairments (such as problems with attention, executive functions, memory and language abilities) are common in people with brain metastases as a result of disease and/or treatment effects. These impairments can significantly limit functional independence, participation in valued roles and activities, and overall quality of life.

Building on research in other cognitively-impaired populations, we designed a brief, structured, patient-centered Cognitive Support Program (CSP) for brain metastases patients, who have the option of participating with a caregiver. Program contents include supportive psychoeducation, mindfulness practice, and strategy training (e.g., strategies to improve memory or concentration). This prospective, single-arm study will enroll 24 brain metastases patients to evaluate the feasibility and preliminary efficacy of the CSP. A battery of outcome measures is administered (1) prior to intervention, (2) after completing the CSP, and (3) after an additional 3 months to evaluate longer-term outcomes. Feasibility assessment will include program retention and adherence. Reliable change analyses will examine treatment effects, with regression analyses to explore moderating effects of select patient, disease and treatment factors (e.g., severity of baseline cognitive impairment, number of brain lesions, cranial radiation dose and distribution). Results of this trial will inform further development and implementation of evidence-based supportive care for cognitively-impaired brain metastases patients.

ELIGIBILITY:
Inclusion Criteria:

* age 18 or older
* able to provide informed consent to all procedures
* diagnosis of one or more brain metastases, with primary cancer outside the CNS
* indication of cognitive deficits from self-report and/or cognitive testing
* interest in participating in a cognitive rehabilitation program
* able to complete study activities

Exclusion Criteria:

* concurrent non-cancer-related neurological or major psychiatric disorder or other medical condition suspected to influence cognition

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-11-28 (Actual); Study Completion 2018-11-28 (Actual)

PRIMARY OUTCOMES:
Functional Assessment of Cancer Therapy - Cognitive | Baseline; 2 months (0-2 weeks post-training); 5 months (3 months post-training)
  Multi-domain cognitive symptom questionnaire completed at each time point. Raw scores are converted to z-scores (M = 0, SD = 1, higher scores = better functioning) according to published criteria, and change from baseline to post-training and to 3-month follow-up calculated by subtraction.

SECONDARY OUTCOMES:
Frontal Systems Behavior Scale | Baseline; 2 months (0-2 weeks post-training); 5 months (3 months post-training)
  Executive cognitive symptom questionnaire completed at each time point. Raw scores are converted to z-scores (M = 0, SD = 1, higher scores = better functioning) according to published criteria, and change from baseline to post-training and to 3-month follow-up calculated by subtraction.
Hopkins Verbal Learning Test - Revised | Baseline; 2 months (0-2 weeks post-training); 5 months (3 months post-training)
  Neurocognitive test of memory completed at each time point. Raw scores are converted to z-scores (M = 0, SD = 1, higher scores = better functioning) according to published criteria, and change from baseline to post-training and to 3-month follow-up calculated by subtraction.
Trail Making Test | Baseline; 2 months (0-2 weeks post-training); 5 months (3 months post-training)
  Neurocognitive test of processing speed and executive function completed at each time point. Raw scores are converted to z-scores (M = 0, SD = 1, higher scores = better functioning) according to published criteria, and change from baseline to post-training and to 3-month follow-up calculated by subtraction.
Wechsler Digit Span Test | Baseline; 2 months (0-2 weeks post-training); 5 months (3 months post-training)
  Neurocognitive test of working memory completed at each time point. Raw scores are converted to z-scores (M = 0, SD = 1, higher scores = better functioning) according to published criteria, and change from baseline to post-training and to 3-month follow-up calculated by subtraction.
BADS Zoo Map Test | Baseline; 2 months (0-2 weeks post-training); 5 months (3 months post-training)
  Neurocognitive test of executive function completed at each time point. Raw scores are converted to z-scores (M = 0, SD = 1, higher scores = better functioning) according to published criteria, and change from baseline to post-training and to 3-month follow-up calculated by subtraction.
Controlled Oral Word Association Test | Baseline; 2 months (0-2 weeks post-training); 5 months (3 months post-training)
  Neurocognitive test of verbal fluency completed at each time point. Raw scores are converted to z-scores (M = 0, SD = 1, higher scores = better functioning) according to published criteria, and change from baseline to post-training and to 3-month follow-up calculated by subtraction.
Functional Assessment of Cancer Therapy - Brain | Baseline; 2 months (0-2 weeks post-training); 5 months (3 months post-training)
  Health-related quality of life questionnaire completed at each time point. Raw scores are converted to z-scores (M = 0, SD = 1, higher scores = better functioning) according to published criteria, and change from baseline to post-training and to 3-month follow-up calculated by subtraction.
Positive and Negative Affect Schedule | Baseline; 2 months (0-2 weeks post-training); 5 months (3 months post-training)
  Quality of life (well-being) questionnaire completed at each time point. Raw scores are converted to z-scores (M = 0, SD = 1, higher scores = better functioning) according to published criteria, and change from baseline to post-training and to 3-month follow-up calculated by subtraction.
Hospital Anxiety and Depression Scale | Baseline; 2 months (0-2 weeks post-training); 5 months (3 months post-training)
  Quality of life (psychological distress) questionnaire completed at each time point. Raw scores are converted to z-scores (M = 0, SD = 1, higher scores = better functioning) according to published criteria, and change from baseline to post-training and to 3-month follow-up calculated by subtraction.
Illness Intrusiveness Rating Scale | Baseline; 2 months (0-2 weeks post-training); 5 months (3 months post-training)
  Quality of life (activity participation) questionnaire completed at each time point. Raw scores are converted to z-scores (M = 0, SD = 1, higher scores = better functioning) according to published criteria, and change from baseline to post-training and to 3-month follow-up calculated by subtraction.

CONTACTS AND LOCATIONS:
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No